CLINICAL TRIAL: NCT04026932
Title: The Clinical Effects of Modified Tinnitus Relieving Sound Treatment
Brief Title: The Clinical Effects of Modified TRS Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Tinnitus sound therapy RCT
Record Dates: First submitted 2019-07-11; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Tinnitus, Subjective
Keywords: subjective tinnitus; tinnitus relieving sound; clinical effects
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unmodified music group (Placebo Comparator): 34 participants in Group 1 will listen to the music without any modification for at least two hours a day in total.
  Interventions: Other: Listening to unmodified music
- Modified tinnitus relieving sound group (Experimental): 34 participants in Group 2 will listen to the music modified according to the matched dominant tinnitus pitch for at least two hours a day in total.
  Interventions: Other: Listening to modified tinnitus relieving sound

INTERVENTIONS:
Other: Listening to unmodified music — Listening to unmodified music for at least 2 hours a day
  Arms: Unmodified music group
Other: Listening to modified tinnitus relieving sound — Listening to modified tinnitus relieving sound for at least 2 hours a day
  Arms: Modified tinnitus relieving sound group

SUMMARY:
Objective Tinnitus is one of the most common acoustic disorders by affecting 5-43% people around the world, and tinnitus is harmful to social and individuals, inducing to annoyance, irritability, anxiety, depression, insomnia and concentration difficulties. Many efforts have been made to help tinnitus suffers, however, the curative means are still in absence. This study aims to introduce a novel sound therapy for tinnitus and to evaluate the efficacy of modified tinnitus relieving sound treatment in comparison with unmodified music which served as a control.

Methods and analysis A randomized, triple-blinded, controlled, clinical trial will be carried out. 68 patients with subjective tinnitus will be recruited and randomized into two groups in 1:1 ratio. The primary outcomes will be Tinnitus Handicapped Inventory (THI), Hospital Anxiety and Distress Scale (HADS), and visual analogue scale (VAS) for tinnitus; the secondary outcome measures will be Athens Insomnia Scale (AIS), tinnitus loudness matched by sensation level (LM, SL), and minimum masking level (MML). Assessment will be performed at baseline and at 1, 3, 9, and 12 months post-randomization. The sound stimulus will be persistent until 9 months after randomization, and be interdictory in the last three months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18 to 80 years old;
2. Diagnosed with subjective tinnitus;
3. Chronic tinnitus: tinnitus course ≥3 months;
4. Be able to understand and communicate with Mandarin；
5. The average pure tone threshold (0.5, 1, 2kHz) ≤ 55dB HL of the worse ear;
6. Subjects are able to understand the purpose of the study, volunteer to participate and cooperate with the instructors to complete the experiment, and be willing to sign the informed consent.

Exclusion Criteria:

1. Pulsatile tinnitus and objective tinnitus；
2. Having significant health issues that affect or prevent participation or continue with the follow-up;
3. Diseases requiring other medical intervention first (eg, infections, tumors, otosclerosis, Meniere's disease, the acute stage of sudden sensorineural hearing loss);
4. People with severe hyperacusis, severe anxiety, depression and other psychiatric disorders；
5. Currently participating in other research projects that may affect tinnitus；
6. Subjects who are not considered suitable for this clinical trial by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicapped Inventory (THI) | 1 months from baseline
  THI is a self-assessment inventory including 25 items with grades four categories of tinnitus severity: slight corresponding to a score 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus.
Tinnitus Handicapped Inventory (THI) | 3 months from baseline
  THI is a self-assessment inventory including 25 items with grades four categories of tinnitus severity: slight corresponding to a score 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus.
Tinnitus Handicapped Inventory (THI) | 9 months from baseline
  THI is a self-assessment inventory including 25 items with grades four categories of tinnitus severity: slight corresponding to a score 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus.
Tinnitus Handicapped Inventory (THI) | 12 months from baseline
  THI is a self-assessment inventory including 25 items with grades four categories of tinnitus severity: slight corresponding to a score 0-16, mild (18-36), moderate (38-56), severe (58-100). The higher the score the more severe the tinnitus.
Hospital Anxiety and Distress Scale (HADS) | 1 months from baseline
  HADS includes two subscales for anxiety and depression, each with respective 7 items, and the grades are valued by scoring: negative (0-7), positive (8-21).
Hospital Anxiety and Distress Scale (HADS) | 3 months from baseline
  HADS includes two subscales for anxiety and depression, each with respective 7 items, and the grades are valued by scoring: negative (0-7), positive (8-21).
Hospital Anxiety and Distress Scale (HADS) | 9 months from baseline
  HADS includes two subscales for anxiety and depression, each with respective 7 items, and the grades are valued by scoring: negative (0-7), positive (8-21).
Hospital Anxiety and Distress Scale (HADS) | 12 months from baseline
  HADS includes two subscales for anxiety and depression, each with respective 7 items, and the grades are valued by scoring: negative (0-7), positive (8-21).
Visual Analogue Scale (VAS) for tinnitus | 1 months from baseline
  Visual Analogue Scale (VAS) for tinnitus is a universal psychometric scale evaluating subjective tinnintus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.
Visual Analogue Scale (VAS) for tinnitus | 3 months from baseline
  Visual Analogue Scale (VAS) for tinnitus is a universal psychometric scale evaluating subjective tinnintus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.
Visual Analogue Scale (VAS) for tinnitus | 9 months from baseline
  Visual Analogue Scale (VAS) for tinnitus is a universal psychometric scale evaluating subjective tinnintus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.
Visual Analogue Scale (VAS) for tinnitus | 12 months from baseline
  Visual Analogue Scale (VAS) for tinnitus is a universal psychometric scale evaluating subjective tinnintus. A total score is 10, from 0 to 10. The higher the score, the more severe the symptom.

SECONDARY OUTCOMES:
Athens Insomnia Scale (AIS) | 1 months from baseline
  AIS grades three categories of sleep disorder: no insomnia scoring below 4, suspicious (4-6), insomnia (7-24)
Athens Insomnia Scale (AIS) | 3 months from baseline
  AIS grades three categories of sleep disorder: no insomnia scoring below 4, suspicious (4-6), insomnia (7-24)
Athens Insomnia Scale (AIS) | 9 months from baseline
  AIS grades three categories of sleep disorder: no insomnia scoring below 4, suspicious (4-6), insomnia (7-24)
Athens Insomnia Scale (AIS) | 12 months from baseline
  AIS grades three categories of sleep disorder: no insomnia scoring below 4, suspicious (4-6), insomnia (7-24)
tinnitus loudness matched by sensation level (LM, SL) | 1 months from baseline
  The loudness of tinnitus is reflected in sensation level (dB SL). Sensation level is defined as the loudness value above hearing threshold at the pitch of tinnitus.
tinnitus loudness matched by sensation level (LM, SL) | 3 months from baseline
  The loudness of tinnitus is reflected in sensation level (dB SL). Sensation level is defined as the loudness value above hearing threshold at the pitch of tinnitus.
tinnitus loudness matched by sensation level (LM, SL) | 9 months from baseline
  The loudness of tinnitus is reflected in sensation level (dB SL). Sensation level is defined as the loudness value above hearing threshold at the pitch of tinnitus.
tinnitus loudness matched by sensation level (LM, SL) | 12 months from baseline
  The loudness of tinnitus is reflected in sensation level (dB SL). Sensation level is defined as the loudness value above hearing threshold at the pitch of tinnitus.
minimum masking level (MML) | 1 months from baseline
  MML test is presented bilaterally, the noise is raised until tinnitus is just covered in both ears. The higher the value, the more severe the tinnitus.
minimum masking level (MML) | 3 months from baseline
  MML test is presented bilaterally, the noise is raised until tinnitus is just covered in both ears. The higher the value, the more severe the tinnitus.
minimum masking level (MML) | 9 months from baseline
  MML test is presented bilaterally, the noise is raised until tinnitus is just covered in both ears. The higher the value, the more severe the tinnitus.
minimum masking level (MML) | 12 months from baseline
  MML test is presented bilaterally, the noise is raised until tinnitus is just covered in both ears. The higher the value, the more severe the tinnitus.

CONTACTS AND LOCATIONS:
Overall Officials: Huawei Li, Study Chair — Eye and ENT Hospital of Fudan University
Locations (1):
- Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langguth B, Kreuzer PM, Kleinjung T, De Ridder D. Tinnitus: causes and clinical management. Lancet Neurol. 2013 Sep;12(9):920-930. doi: 10.1016/S1474-4422(13)70160-1. PMID 23948178
- [Background] De Ridder D, Elgoyhen AB, Romo R, Langguth B. Phantom percepts: tinnitus and pain as persisting aversive memory networks. Proc Natl Acad Sci U S A. 2011 May 17;108(20):8075-80. doi: 10.1073/pnas.1018466108. Epub 2011 Apr 18. PMID 21502503
- [Background] Tunkel DE, Bauer CA, Sun GH, Rosenfeld RM, Chandrasekhar SS, Cunningham ER Jr, Archer SM, Blakley BW, Carter JM, Granieri EC, Henry JA, Hollingsworth D, Khan FA, Mitchell S, Monfared A, Newman CW, Omole FS, Phillips CD, Robinson SK, Taw MB, Tyler RS, Waguespack R, Whamond EJ. Clinical practice guideline: tinnitus. Otolaryngol Head Neck Surg. 2014 Oct;151(2 Suppl):S1-S40. doi: 10.1177/0194599814545325. PMID 25273878
- [Background] Cima RF, Maes IH, Joore MA, Scheyen DJ, El Refaie A, Baguley DM, Anteunis LJ, van Breukelen GJ, Vlaeyen JW. Specialised treatment based on cognitive behaviour therapy versus usual care for tinnitus: a randomised controlled trial. Lancet. 2012 May 26;379(9830):1951-9. doi: 10.1016/S0140-6736(12)60469-3. PMID 22633033
- [Background] Newman CW, Jacobson GP, Spitzer JB. Development of the Tinnitus Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1996 Feb;122(2):143-8. doi: 10.1001/archotol.1996.01890140029007. PMID 8630207
- [Derived] Tang D, Wang J, Yu X, Yu H. The clinical effects of modified tinnitus relieving sound (MTRS) for chronic tinnitus: protocol for a randomized controlled trial. Trials. 2023 Jun 2;24(1):372. doi: 10.1186/s13063-023-07389-8. PMID 37268971